CLINICAL TRIAL: NCT07346443
Title: Mechanism Study of G Protein-coupled Receptor 81 in Multiple Organ Dysfunction of Heat Stroke
Status: Not yet recruiting | Type: Observational
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: SAHoWMU-CR2025-03-136
Record Dates: First submitted 2026-01-05; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Heat Stroke
Keywords: G protein-coupled receptor 81; Lactic Acid; heat stroke
MeSH Terms: conditions — Heat Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- heatstroke group: heatstroke patient, no intervention

SUMMARY:
Heat stroke is one of the common acute and critical conditions in the ICU, characterized by a high incidence and mortality rate, and there is still a lack of effective and precise treatment methods. The latest research indicates that G protein-coupled receptor 81 (GPR81), as an endogenous receptor of lactic acid, can regulate immune responses by up-regulating the expression of inflammatory factors and the chemotaxis of neutrophils, suggesting that the GPR81 receptor may play a potential key role in heat stroke. The investigators aim to reveal the position and key role of GPR81 in improving multiple organ dysfunction caused by heat stroke, and to clarify its specific molecular mechanism, with the goal of providing new ideas for the prevention and treatment of heat stroke based on lactate levels, a commonly used clinical indicator.

ELIGIBILITY:
Inclusion Criteria:

* 1) There was a clear history of high-temperature exposure before the onset of the disease; 2) Core body temperature ≥40℃ upon admission or within 2 hours of onset; 3) At least one abnormal symptom of the central nervous system occurs 4) Sign an informed consent form or have their legal representative agree to participate in the research.

Exclusion Criteria:

* 1) Suffering from central nervous system diseases; 2) Long-term use of anticoagulants; 3) Those who refuse to participate or withdraw their informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients who are diagnosed with heatstroke
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
The 28-day survival rate of patients with heat stroke | Survival status will be assessed over a period of up to 28 days, starting from the date of hospital admission.
  For patients with heat stroke, if they die within 28 days, it indicates they are non-survivors; if they do not die within 28 days, it indicates they are survivors

SECONDARY OUTCOMES:
Plasma lactate levels in patients with heat stroke | Plasma lactate levels will be measured at admission and then daily during the hospital stay, for a period of up to 28 days.
  Collect the plasma lactic acid level each time when patients with heat stroke are hospitalized

IPD SHARING:
Plan to Share IPD: Yes
Study protocol and statistical analysis plan.
Supporting Information: SAP
Time Frame: Beginning 6 months after publication with no end date
Access Criteria: Deidentifed participant data underlying the findings wil be made available upon reasonable request. proposls fordata acess should be directedto the corresponding author Shengwei Jin
URL: https://www.wzhealth.com/